CLINICAL TRIAL: NCT02859272
Title: Vaginal Vault Suspension During Benign Hysterectomy. A Questionnaire and Register-based Study.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nykøbing Falster County Hospital (Other)
Collaborators: Zealand University Hospital (Other); Copenhagen University Hospital, Denmark (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Lisbeth Bonde, M.D., Research Fellow, Nykøbing Falster County Hospital
Other Study IDs: REG-30-2013
Record Dates: First submitted 2016-07-15; First posted 2016-08-09 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Postoperative Pelvic Organ Prolapse; Benign Hysterectomy; Suspension
Keywords: Suspension, benign hysterectomy, post operative prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Female pelvic organ prolapse (POP) is characterized by lack of vaginal support which enables pelvic organs to bulge into the vaginal walls and sometimes protrude through the genital hiatus. POP is more frequent among women who had their uterus removed.

We would like to investigate whether suspension of the top of the vagina during remowal of the uterus prevents subsequent POP.

The purpose of the PhD project is therefore to describe validity, terminology, and operative performance of used suspension methods during benign hysterectomy in Denmark. Further, to investigate these suspension methods' possible association with pain, life quality, sexuality, pessary use, and POP .

DETAILED DESCRIPTION:
In 2012 the investigators introduced codes of suspension methods to the Danish hysterectomy and hysteroscopy Database's registration chart. Consequently, validity of these codes needs to be ensured to enable their use in further research.

Thereafter, the prevalence of Danish gynecologists' use of the different suspension methods will be investigated. A questionnaire will elucidate a possible relation between the suspension methods and pain, life quality and sexuality. Through a register based study in the National Patient Register the association between suspension methods and post hysterectomy POP and possible confounding will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Alive women two years after hysterectomy
* Benign hysterectomy
* Willingness to participate (in the questionnaire)

Exclusion Criteria:

* Death
* Emigration
* Secret address

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women operated with a benign hysterectomy from May 2012-June 2014.
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Through national registries investigate the prevalence of postoperative pelvic organ prolapse among hysterectomized women in relation to performed suspension method. | 6 months

SECONDARY OUTCOMES:
Through a questionnaire investigate postoperative pain in relation to suspension method. | 2 years
Through a questionnaire investigate life quality in relation to suspension method. | 2 years
Through a questionnaire investigate sexuality in relation to suspension method. | 2 years
Validity of suspension methods | 6 months
  Assessment of agreement between the description of suspension method in 600 medical records of hysterectomy and the corresponding registration of suspension methods in the Danish Hysterectomy and hysteroscopy database.